CLINICAL TRIAL: NCT01169324
Title: Effect of DBS on Sleep Architecture in Patients With Movement Disorders.
Brief Title: Effect of Deep Brain Stimulation (DBS) on Sleep Architecture in Patients With Movement Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Amy Amara, MD, Instructor, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: F100528004
Record Dates: First submitted 2010-07-02; First posted 2010-07-26 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Parkinson's Disease; Tremor; Dystonia
Keywords: Parkinson's disease; Tremor; Dystonia; DBS; Sleep
MeSH Terms: conditions — Parkinson Disease; Tremor; Dystonia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DBS on (Experimental): baseline settings
  Interventions: Other: Alteration of DBS stimulator settings
- DBS off (No Intervention): DBS off

INTERVENTIONS:
Other: Alteration of DBS stimulator settings — Alteration of DBS stimulator settings
  Arms: DBS on

SUMMARY:
The purpose of this prospective, participant-blinded trial is to determine the changes in sleep architecture in a cohort of subjects who have undergone deep brain stimulation (DBS) surgery for treatment of movement disorders such as moderate to advanced Parkinson's disease (PD), tremor, or dystonia. Our preliminary observational data suggest that unilateral subthalamic nucleus (STN) DBS improves subjective sleep quality in PD patients 6 months after the procedure. The cause of this improvement in sleep quality is unknown, and this study proposes the use of polysomnography (PSG) to test whether the improvement in sleep is independent of improvement in night-time mobility associated with DBS treatment of the motor symptoms of PD, tremor, or dystonia.

ELIGIBILITY:
Inclusion Criteria:

* Prior DBS surgery for treatment of movement disorders such as PD, tremor, or dystonia.
* Stable DBS stimulator settings and medication regimen for at least 6 weeks prior to the sleep studies.
* Sleep dysfunction as measured by the Pittsburgh Sleep Quality Index (PSQI) (score >5) at the subject's baseline pre-surgical evaluation.

Exclusion Criteria:

* Known narcolepsy
* Other previous surgical treatment of Parkinson's disease, tremor, or dystonia (with the exception of DBS) including pallidotomy, thalamotomy, or gene therapy procedures.
* Untreated obstructive sleep apnea. If obstructive sleep apnea is discovered during the first sleep study, the subject will be removed from the study. After they have been treated for at least 6 weeks with CPAP, they can re-start the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-07-15 (Actual); Primary Completion 2015-12-11 (Actual); Study Completion 2015-12-11 (Actual)

PRIMARY OUTCOMES:
Sleep Efficiency | 1 month
  This is the percentage of time the subject is in bed when he/she is actually asleep.

SECONDARY OUTCOMES:
Wake after sleep onset (WASO) | 1 month
  This is a measurement of the amount of time during polysomnography recording that the subject is awake after their initial sleep onset.
Total Sleep Time | 1 month
Two timed motor tasks | 1 month
  1. The subject will tap index finger between 2 points 30 cm apart on the table for 10 seconds.
  2. The subject will be timed as they rise from a chair, walk 7 meters, return to the chair, and sit down.

CONTACTS AND LOCATIONS:
Overall Officials: Amy W Amara, MD, phD, Principal Investigator — UAB Neurology
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States